CLINICAL TRIAL: NCT04683536
Title: Bakircay University Cigli Training and Research Hospital
Acronym: BUCEAH
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Ozan HORSANALI, Bakircay University Cigli Training and Research Hospital, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: Cigli
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Bladder Cancer
Keywords: obturator nerve blockade; bladder cancer; non-muscle invasive bladder cancer; adductor contraction; bladder perforation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Patients underwent TUR-BT under spinal anesthesia
  Interventions: Procedure: Obturator nerve blockade
- Study group: Patients underwent TUR-BT under spinal anesthesia combined with ultrasound guided obturator nerve blockade
  Interventions: Procedure: Obturator nerve blockade

INTERVENTIONS:
Procedure: Obturator nerve blockade — We performed spinal anesthesia combined with ultrasound guided obturator nerve blockade according to the localization of bladder cancer in patients with lateral wall localized non-muscle invasive bladder cancer

SUMMARY:
The aim of the study is to investigate the oncological outcomes of obturator nerve blockade in patients with lateral wall localized non-muscle invasive bladder cancer

DETAILED DESCRIPTION:
Patient divided into two group.First group includes patients underwent TUR-BT under only spinal anesthesia and second group includes patients underwent TUR-BT under spinal anesthesia combined with ultrasound guided obturator nerve blockade.

ELIGIBILITY:
Inclusion Criteria:

* patients with lateral wall localized non muscle invasive bladder cancer

Exclusion Criteria:

* history of previous TUR-BT
* diagnosis of non-urothelial carcinoma
* coagulopathy
* history of allergic reaction to the local anesthtetic agent
* presence of muscle-invasive bladder cancer
* history of chemotherapy or radiotherapy before TUR-BT
* precence of variant histopathology
* using bipolar energy for the resection of bladder tumor
* presence of concomittant upper urothelial tract urothelial carcinoma
* patients with the neuromusculer disease
* pregnancy
* history of medication effecting immune system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with lateral wall localized non muscle invasive bladder cancer underwent TUR-BT under spinal anesthesia combined with ultrasound guided obturator nerve blockade
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Oncological outcomes | 5 year
  Reccurens or progression of tumor was recorded

SECONDARY OUTCOMES:
Complications | 5 years
  Complications during surgery was recorded

IPD SHARING:
Plan to Share IPD: No